CLINICAL TRIAL: NCT07058636
Title: Evaluation of the Efficacy of Adding Greater Occipital Nerve Block to Trigger Point Injection in Patients With Neck Pain and Upper Trapezius Trigger Points: A Single-Blind Randomized Controlled Trial
Brief Title: Efficacy of Adding Greater Occipital Nerve Block to Trigger Point Injection in Patients With Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Başak Mansız-Kaplan, Principal İnvestigator ,specialist doctor, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEŞH-EK-2025-013
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain; Myofacial Pain Syndrome; Trigger Point Pain, Myofascial; Trigger Points; Upper Trapezius Trigger Points; Cervicogenic Headache
Keywords: neck pain; myofascial pain syndrome; trigger point injection; ultrasound guided occipital nerve block; upper trapezius trigger point
MeSH Terms: conditions — Neck Pain; Facial Neuralgia; Myofascial Pain Syndromes; Post-Traumatic Headache | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Our study was designed as a prospective, single-blind, randomized controlled trial. Patients who presented to the PMR outpatient clinic and were diagnosed with myofascial pain syndrome will be included in the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trigger Point Injection Group (Active Comparator): Patients in this arm will receive trigger point injections only. The injection solution consists of 1 ml of 2% lidocaine mixed with 1 ml of normal saline
  Interventions: Drug: 2% Lidocaine HCl + saline
- Trigger Point Injection Plus Ultrasound-Guided Greater Occipital Nerve Block Group (Active Comparator): Patients in this arm will receive the same trigger point injection protocol plus an ultrasound-guided greater occipital nerve (GON) block. The GON block solution consists of a mixture of 1 ml of 2% lidocaine, and 1 ml of betamethasone.
  Interventions: Drug: 2% Lidocaine HCl + saline; Drug: Steroid+lidocaine

INTERVENTIONS:
Drug: 2% Lidocaine HCl + saline — The intervention consists of injecting a mixture of 1 ml 2% lidocaine and 1 ml normal saline into trigger points located in the upper trapezius muscle.
Drug: Steroid+lidocaine — The GON block involves injecting a mixture of 1 ml 2% lidocaine and 1 ml betamethasone.
  Arms: Trigger Point Injection Plus Ultrasound-Guided Greater Occipital Nerve Block Group

SUMMARY:
Study Title:

Evaluation of the Effectiveness of Adding Greater Occipital Nerve Block to Trigger Point Injection in Patients with Neck Pain Due to Upper Trapezius Trigger Points: A Single-Blind Randomized Controlled Trial

Purpose of the Study:

This study aims to evaluate whether adding a Greater Occipital Nerve (GON) block to the standard trigger point injection treatment provides better pain relief and improves daily function in patients with neck pain caused by trigger points in the upper trapezius muscle. Trigger points are small, sensitive spots in muscles that can cause significant pain and discomfort. While both trigger point injections and GON blocks are common treatments for neck and head pain, it is not yet clear if combining these two methods offers better results.

Why is this study important? Neck pain related to trigger points in the upper trapezius muscle is a frequent problem, but there is limited research on the effectiveness of combining trigger point injections with GON blocks. This study will provide important information on whether the combination therapy can reduce pain more effectively and improve patients' quality of life and ability to perform daily activities.

Who can participate?

Adults aged 18 to 65 years old

Diagnosed with myofascial pain syndrome (MAS) based on specific clinical criteria, including the presence of trigger points in the upper trapezius muscle

Experiencing neck pain lasting longer than 3 months

Pain intensity rated 5 or higher on a scale of 0 to 10

Who cannot participate?

Pregnant or breastfeeding women, children, elderly people, unconscious or critically ill patients

Patients with allergies to local anesthetics or steroids

Individuals with bleeding disorders or infections near the injection site

Patients with serious psychiatric or neurological diseases, or other medical conditions that may affect study results

Those who have recently received similar treatments or surgery for neck or shoulder problems

Study Design and Procedures:

The study will include 60 patients meeting the criteria, randomly assigned to two groups using a balanced randomization method.

Group A will receive only trigger point injections into the upper trapezius muscle using a mixture of lidocaine and saline solution.

Group B will receive both trigger point injections and an ultrasound-guided GON block, which involves injecting a combination of local anesthetics and steroid near the greater occipital nerve to reduce pain signals.

Both groups will receive the same home exercise program focusing on stretching and strengthening neck muscles to support recovery. Patients will be encouraged to perform these exercises regularly and will be followed up weekly by phone to check their progress.

The doctor assessing patients' progress will not know which treatment the patient received, to ensure unbiased results.

Assessments:

Patients will be evaluated at three different times: before treatment, 1 week after treatment, and 4 weeks after treatment. Assessments include:

Pain intensity and quality (using Visual Analog Scale and McGill Pain Questionnaire)

Neck disability and ability to perform daily activities (Neck Disability Index)

Quality of life (Nottingham Health Profile)

Neck joint movement and position sense (using clinical tests with special equipment)

Posture evaluation (measuring head position using photography)

Expected Outcomes:

The main goal is to determine if the combined treatment of trigger point injection plus GON block is more effective than trigger point injection alone in reducing pain, improving neck function, and enhancing quality of life.

Duration and Follow-Up:

The study is planned to last 12 months. Patients will be closely monitored during and after treatment to ensure safety and to collect necessary data.

Potential Benefits and Risks:

Participants may experience pain relief and improved function if the combined treatment is effective. Risks include mild discomfort or side effects related to injections, which will be minimized by experienced medical staff.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years.
* Diagnosed with myofascial pain syndrome (MPS) based on the major and minor criteria described by Travell and Simons (a diagnosis requires all 5 major and at least 1 minor criterion)
* Presence of active trigger points in the upper trapezius muscle.
* Patients with neck pain lasting longer than 3 months.
* Pain intensity of ≥5 on the Visual Analog Scale (VAS).

Exclusion Criteria:

* Elderly, pediatric, pregnant, postpartum, or breastfeeding individuals; patients in intensive care; unconscious individuals; or legally incapacitated persons.
* Known allergy to local anesthetics used in trigger point injection (e.g., lidocaine, bupivacaine) or to other drugs used (e.g., corticosteroids).
* Patients with bleeding disorders (e.g., hemophilia, thrombocytopenia) or those currently on anticoagulant therapy.
* Presence of active infection at or near the injection site, or any systemic infection; impaired skin integrity.
* Patients with psychiatric disorders that may interfere with treatment response or affect study outcomes.
* Patients with severe neurological or cardiovascular disorders, or with uncontrolled diabetes.
* Patients with cervical disc pathologies with radiculopathy.
* History of receiving shoulder injection, trigger point injection, dry needling, manual therapy, or electrotherapy within the past 3 months.
* History of cervical or shoulder surgery.
* Patients diagnosed with adhesive capsulitis, rotator cuff tendinopathy, or shoulder impingement syndrome.
* Diagnosis of fibromyalgia.
* Presence of active trigger points in other back muscles.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, Week 1 and Week 4 post-intervention.
  Global pain assessment using a Visual Analog Scale ranging from 0 ("no pain") to 10 ("unbearable pain"). Patients rate their pain intensity on this scale.

SECONDARY OUTCOMES:
McGill-Melzack Pain Questionnaire | Baseline, Week 1 and Week 4 post-intervention.
  A tool assessing qualitative and quantitative aspects of pain, including sensory, affective, and overall pain components.
Neck Disability Index (NDI) | Baseline, Week 1, and Week 4 post-intervention.
  A 10-item questionnaire evaluating functional limitations and disability caused by neck pain in daily activities.
Nottingham Health Profile (NHP) | Baseline, Week 1 and Week 4 post-intervention.
  A patient-reported questionnaire measuring subjective health status and quality of life across six dimensions: energy, pain, emotional reactions, sleep, social isolation, and physical mobility.
Cervical Joint Position Error Test (Proprioception Assessment) | Baseline, Week 1 and Week 4 post-intervention.
  Measurement of cervical proprioception errors during head and neck movements using a laser pointer and target board system. The average error in centimeters over six repetitions per movement will be recorded.
Cervical Range of Motion (CROM) Measurement | Baseline, Week 1 and Week 4 post-intervention.
  Objective measurement of cervical spine active range of motion in degrees using a goniometer.

OTHER OUTCOMES:
Craniovertebral Angle Measurement | Baseline only
  Assessment of forward head posture using photogrammetric measurement of the craniovertebral angle. The angle is formed between a horizontal line passing through the C7 spinous process and a line connecting the tragus of the ear to C7. Smaller angles indicate a more pronounced forward head posture.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No